CLINICAL TRIAL: NCT04215081
Title: ExoAtlet II Lower Extremity Exoskeleton Safety and Efficacy Use With Spinal Cord Injured Individuals
Brief Title: ExoAtlet II For SCI Patients
Acronym: EXOATLET2SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: COSMO ROBOTICS CO., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EA22019SCI
Record Dates: First submitted 2019-12-20; First posted 2020-01-02 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Spinal Cord Injuries; Paraplegia
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia

STUDY DESIGN:
Intervention Model Description: SCI Level T4-L5 or, C7-T3 with ASIA D
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ExoAtlet II Safety and Efficacy (Experimental): 20 participants with paraplegia from SCI will participate in gait training using ExoAtlet II powered exoskeleton.
  Interventions: Device: Gait training using ExoAtlet exoskeleton

INTERVENTIONS:
Device: Gait training using ExoAtlet exoskeleton — Subjects will learn to use the ExoAtlet II exoskeleton, with the assistance of a trained medical professional, to perform functional activities (including stand-up, sit-down, stepping forward, and walking).

SUMMARY:
This study will evaluate the ExoAtlet II exoskeleton for safety and effectiveness of providing persons with a spinal cord injury (SCI) who are non-ambulatory or have limited ambulatory function, to stand up and ambulate under a variety of conditions.

DETAILED DESCRIPTION:
The study will introduce the ExoAtlet II exoskeleton to SCI patients with lower extremity paralysis (partial or complete) and provide rehabilitative standing and walking intervention. The study will be conducted with a trained clinician that will fit each patient into the adjustable exoskeleton system and provide customized programming to meet each user's specific needs. The training program will be initiated based upon each patient's comfort in the exoskeleton and ability to stand with assistance. Each patient will be closely monitored to assess ongoing health as well as their individual standing and walking ability. All exoskeleton sessions will be performed with a trained medical professional controlling the exoskeleton. Patient safety is the primary concern and all adverse events will be documented and addressed. This study will evaluate the ExoAtlet 2.0 exoskeleton for safety and effectiveness of providing persons with a spinal cord injury (SCI) who are non-ambulatory or have limited ambulatory function, the ability to stand up and walk in a clinical facility.

ELIGIBILITY:
Inclusion Criteria:

1. 18 Years of age or older in general good health
2. Weight, no more than 220lbs (100kg)
3. Skin must be healthy where it touches the ExoAtlet 2.0
4. Able to stand using a device such as a standing frame
5. Have enough strength in your hands and shoulders to support yourself standing and walking using crutches or a walker
6. Have good control of upper body
7. Determined to have enough bone health to walk full weight bearing without risk of fracture. Meeting of this condition is at the discretion of your personal MD
8. Passive range of motion (PROM) at shoulders, trunk, upper extremities and lower extremities within functional limits for safe gait and use of appropriate assistive device/stability aid
9. Hip width no greater than 18" (46 cm) measured when sitting.
10. Femur length between 37 cm and 49 cm measured between mid patellar tendon and the floor.
11. In general, good health and able to tolerate moderate levels of activity.
12. Blood pressure and heart rate within established guidelines for locomotive training: At rest; Systolic 150 or less Diastolic 90 or less and Heart rate 100 or less Exercise; Systolic 180 or less, Diastolic 105 or less and Heart Rate 145 or less

Exclusion Criteria:

1. Spinal cord injury level higher than T4 or C7 ASIA D
2. Severe muscle stiffness/tightness
3. Significant spasticity (Modified Ashworth Scale score of 3 or above)
4. Trunk or lower extremity pressure ulcer
5. Open Wounds/tissue hypersensitivity
6. Unstable spine, un-healed limbs, or fractures
7. Severe sensitivity to touch
8. Presence of bone in soft tissue where bone normally does not exist (heterotopic ossification), limiting range of motion in the hip or knee joints
9. Joint instability, dislocation, moderate to severe hip dysplasia
10. Significant scoliosis (>40 degrees)
11. Hardware, implant, or any external device impeding with safe fitting or use of ExoAtlet 2.0
12. Femoral or tibial rotation deformity (>15 degrees)
13. Significant flexion contractures limited to 35º at the hip and 20º at the knee
14. Uncontrolled seizures, musculoskeletal injury, fracture or lower-limb surgery in past year.
15. Known history of pulmonary disease limiting exercise tolerance or history of cardiac disease
16. Psychopathology, or other condition that the physician or investigator, in his or her clinical judgment, considers to be exclusionary to safely use an exoskeleton.
17. Severe concurrent medical diseases, illness, systemic or peripheral infection
18. Dizziness or headache with standing
19. History of autonomic dysreflexia
20. Orthostatic Hypotension: Decrease in Systolic BP > 20, Diastolic BP > 10 upon standing from a seated position.
21. Pregnant or lactating females

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-01-04 (Actual); Study Completion 2020-01-04 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 0-8 weeks
  Document and track any adverse events, both minor and major, during exoskeleton sessions.
Skin integrity | 0-8 weeks
  A visual inspection of the participant's skin, at all areas of contact with the exoskeleton, will be conducted at the beginning and end of each session.

SECONDARY OUTCOMES:
10 Meter Walk Test | 1 Day
  Assesses walking speed, in the exoskeleton, in meters per second over a distance of 10 meters
6 Minute Walk Test | 1 Day
  Record the distance covered during a 6 minute walk test utilizing the exoskeleton, to evaluate users endurance
Transfer in and out | 2 Days
  Percentage of patients able to successfully transfer in and out of the exoskeleton with or without assistance
Perform Sit to Stand to Sit | 2 Days
  Percentage of patients that successfully completed both sit to stand and stand to sit in the exoskeleton

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Kotov, MD, Principal Investigator — Moscow Regional Research and Clinical Institute (MONIKI)
Locations (1):
- Moscow Regional Research Clinical Institute. M.F. Vladimirsky, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gagnon DH, Cunha JD, Boyer-Delestre M, Bosquet L, Duclos C. How does wearable robotic exoskeleton affect overground walking performance measured with the 10-m and six-minute walk tests after a basic locomotor training in healthy individuals? Gait Posture. 2017 Oct;58:340-345. doi: 10.1016/j.gaitpost.2017.08.027. Epub 2017 Aug 26. PMID 28865396
- [Background] Miller LE, Zimmermann AK, Herbert WG. Clinical effectiveness and safety of powered exoskeleton-assisted walking in patients with spinal cord injury: systematic review with meta-analysis. Med Devices (Auckl). 2016 Mar 22;9:455-66. doi: 10.2147/MDER.S103102. eCollection 2016. PMID 27042146
- [Background] Tefertiller C, Hays K, Jones J, Jayaraman A, Hartigan C, Bushnik T, Forrest GF. Initial Outcomes from a Multicenter Study Utilizing the Indego Powered Exoskeleton in Spinal Cord Injury. Top Spinal Cord Inj Rehabil. 2018 Winter;24(1):78-85. doi: 10.1310/sci17-00014. Epub 2017 Nov 20. PMID 29434463
- [Background] Hartigan C, Kandilakis C, Dalley S, Clausen M, Wilson E, Morrison S, Etheridge S, Farris R. Mobility Outcomes Following Five Training Sessions with a Powered Exoskeleton. Top Spinal Cord Inj Rehabil. 2015 Spring;21(2):93-9. doi: 10.1310/sci2102-93. Epub 2015 Apr 12. PMID 26364278
- [Background] Kozlowski AJ, Bryce TN, Dijkers MP. Time and Effort Required by Persons with Spinal Cord Injury to Learn to Use a Powered Exoskeleton for Assisted Walking. Top Spinal Cord Inj Rehabil. 2015 Spring;21(2):110-21. doi: 10.1310/sci2102-110. Epub 2015 Apr 12. PMID 26364280
- [Background] McIntosh K, Charbonneau R, Bensaada Y, Bhatiya U, Ho C. The Safety and Feasibility of Exoskeletal-Assisted Walking in Acute Rehabilitation After Spinal Cord Injury. Arch Phys Med Rehabil. 2020 Jan;101(1):113-120. doi: 10.1016/j.apmr.2019.09.005. Epub 2019 Sep 27. PMID 31568761